CLINICAL TRIAL: NCT04624958
Title: Zanubrutinib and Rituximab Followed by R-DHAOx (Rituximab, Dexamethasone, Cytarabine and Oxaliplatin) Regimen Then Maintenance with Zanubrutinib for Newly-Diagnosed Mantle Cell Lymphoma (MCL): a Single Arm, Open Label, Multi-center Phase II Study
Brief Title: Zanubrutinib and Rituximab Followed by R-DHAOx Then Maintenance with Zanubrutinib for Newly-Diagnosed MCL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-232-01
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Mantle Cell Lymphoma; Newly-diagnosed Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — zanubrutinib; Rituximab; Medicare Part B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- zanubrutinib, rituximab, consolidation chemotherapy and zanubrutinb maintenance (Experimental): Part A (Zanubrutinib and Rituximab): Patients receive zanubrutinib on days 1-28 and rituximab on day 1. Treatment cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity or until patients achieve CR.
  PART B (Consolidation chemotherapy of R-DHAOx): Patients receive R-DHAOx regimen every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Elderly patients (> 65 years old) and patients who achieved CR and minimal residual disease negative after PART B receive zanubrutinb maintenance therapy. Young patients (<65 years old) who achieved CR but minimal residual disease positive after PART B can receive autologous stem cell transplantation and then zanubrutinb maintenance therapy. Patients with PD, SD or PR after PART B quit the trial.
  ZANUBRUTINB MAINTENANCE: Patients receive zanubrutinib every day for up to one year.
  Interventions: Drug: Zanubrutinib and Rituximab; Drug: R-DHAOx; Drug: Zanubrutinib Maintenance

INTERVENTIONS:
Drug: Zanubrutinib and Rituximab — Zanubrutinb 160mg PO BID d1-28; Rituximab 375mg/m2 iv.drip d1.
  Other Names: PART A
Drug: R-DHAOx — Rituximab 375mg/m2 iv.drip d1; Dexamethasone 20mg iv.drip d1-4; Cytarabine 2000mg/m2 (1000mg/m2 for patients aged over 65) iv.drip d2,3 Oxaliplatin 130mg/m2 iv.drip d1.
  Other Names: PART B
Drug: Zanubrutinib Maintenance — Zanubrutinb 160mg PO BID.

SUMMARY:
This phase 2 trial studies the efficacy and safety of zanubrutinib plus rituximab followed by R-DHAOx (rituximab, dexamethasone, cytarabine and oxaliplatin) regimen then maintenance with zanubrutinib for newly-diagnosed Mantle Cell Lymphoma (MCL).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD20 positive mantle cell lymphoma;
* Patients with MCL-related symptomatic and need immediate therapy; Include any of the following: (1) Blastoid variant (2) Pleomorphic variant (3) Ki-67 ≥30% (4) Bulky mass > 7 cm or ≥2 tumors, each ≥5 cm in diameter (5) Mutations in TP53, c-MYC or NOTCH genes (6) Size of spleen ≥20 cm (7) Lymphoma B symptoms (8) Mantle Cell International Prognostic Score (MIPI) > 3 (9) Lymphoma threatening organ function (10) Elevated lactate dehydrogenase (11) Peripheral blood white blood cell > 50×10^9/L (12) Pancytopenia due to bone marrow involvement (13) Pain due to lymphoma;
* Patients received no prior anti-lymphoma treatment;
* At least one evaluable lesion according to 2014 Lugano criteria;
* Ann Arbor stage II-IV;
* Eastern Cooperative Oncology Group (ECOG) of 0-2;
* Life expectancy > 3 months;
* Able to participate in all required study procedures;
* Proper functioning of the major organs: 1) The absolute value of neutrophils (>1.5×10^9/L); 2) platelet count (> 75×10^9/L); 3) Hemoglobin (> 80 g/L); 4) Serum creatinine <1.5 times Upper Limit Normal (ULN) ; 5) Serum total bilirubin < 1.5 times ULN; 6) Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) < 2.5 times ULN; 7) Coagulation function: International Normalized Ratio (INR), Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT) < 1.5 times ULN (unless the subject is receiving anticoagulant therapy and PT and APTT are within the expected range at screening time);

Exclusion Criteria:

* Involvement of central nervous system (CNS)
* Patients with Hemophagocytic syndrome;
* Patients with active bleeding, bleeding tendency or require anticoagulation treatment;
* Patients require treatment with strong CYP3A inhibitors;
* Uncontrolled active infection, with the exception of tumor-related B symptom fever;
* History of human immunodeficiency virus (HIV) infection and/or patients with acquired immunodeficiency syndrome are known;
* Patients with active hepatitis B or active hepatitis C. Patients who are positive for hepatitis B Surface Antigen (HBsAg) or hepatitis C Virus (HCV) antibodies at screening stage must pass further detection of hepatitis B Virus (HBV) DNA (no more than 1000 IU/mL) and HCV RNA (no more than the lower limit of the detection method) in the row. Hepatitis B carriers, stable hepatitis B (DNA titer should not be higher than 1000 IU/mL) after drug treatment, and cured hepatitis C patients can be enrolled in the group;
* Diagnosed with or receiving treatment for malignancy other than lymphoma;
* Pregnant or breastfeeding women;
* Other researchers consider it unsuitable for patients to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate after PART A | 3 years
  Complete remission rate will be determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Complete remission rate after study treatment | 3 years
  Complete remission rate will be determined on the basis of investigator assessments according to 2014 Lugano criteria.
Objective Response rate | 3 years
  Objective Response rate will be determined on the basis of investigator assessments according to 2014 Lugano criteria.
Progression Free Survival | 5 years
  The time from the start of treatment to the progression of the tumor or death (due to any cause).
Overall Survival | 5 years
  The time from the start of treatment to time of death (due to any cause).
Time to Response | 3 years
  The time from the start of treatment to the first assessment of complete remission or partial remission.
Duration of Response | 5 years
  The time from the first assessment of complete remission or partial remission to progressive disease or death (due to any cause).
Percentage of Participants With Adverse Events | 3 years
  Adverse Events will be determined and graded on the basis of investigator assessments according to NCI CTC AE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Qingqing Cai, MD, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong